CLINICAL TRIAL: NCT06746467
Title: the Effect of Vernal Keratoconjunctivitis on Corneal Topographic Profiles
Brief Title: Corneal Topography in Vernal Keratoconjunctivitis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Monica Basem Fayez, assistant lecture, Assiut University
Other Study IDs: corneal topography in vkc
Record Dates: First submitted 2024-12-16; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Keratoconjunctivitis
Keywords: corneal topography on vkc
MeSH Terms: conditions — Keratoconjunctivitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: pentacam — evaluate corneal changes by pentacam

SUMMARY:
To evaluate the corneal topographic changes in VKC patients using Pentacam and prevalence of KC development in VKC.

DETAILED DESCRIPTION:
Vernal keratoconjunctivitis (VKC) is a chronic allergic disease, with seasonal periods of exacerbation.VKC is characterized by itching, photophobia. white mucous discharge, lacrimation, foreign body sensation, and pain due to corneal involvement of shield ulcers. Corneal involvement in VKC involves injury to the superficial and basal epithelial layers and anterior stroma . Excessive eye rubbing and a slow release of matrix metalloproteinases penetrate the cornea in presence of chronic epithelial damage causing astigmatism and corneal ectasia . These changes may be undetected until advanced complications such as keratoconus(KC) with thinning and protrusion of cornea leading to myopia and astigmatism . These changes can be measured accurately by corneal topography, making it the gold standard in the screening of keratoconus and other corneal ectasias . Corneal topography is a method of computer-assisted examination of the cornea in which multiple concentric light rings are projected on cornea. Changes in corneal topography indices to be studied include changes in effective refeactivepower ,asphericity , corneal asymmetry index and visual performance . It is a non-invasive exploratory technique to analyse both qualitatively and quantitatively the morphology of the cornea . The Penta Cam is a cornea and anterior segment topography device, based on a rotating Scheimpflug camera. Its optical cross-sectional analysis that helps in imaging of anterior and posterior corneal surfaces which provides with fullpachymetric map and many other data such as corneal aberrometry and densitometry that allow early detection of ectasia.

ELIGIBILITY:
Inclusion Criteria:

clinical diagnosis of vernal keratoconjunctivitis -

Exclusion Criteria:

patients with corneal disease as corneal opacity, corneal dystrophy or degenerative changes patients with previous corneal surgery patients with ocular trauma.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients will be selected from primary clinic
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
evaluate the corneal topographic changes in VKC patients using Pentacam | 1 year

SECONDARY OUTCOMES:
prevalence of KC development in VKC | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Result] Dantas PE, Alves MR, Nishiwaki-Dantas MC. Topographic corneal changes in patients with vernal keratoconjunctivitis. Arq Bras Oftalmol. 2005 Sep-Oct;68(5):593-8. doi: 10.1590/s0004-27492005000500004. Epub 2005 Nov 28. PMID 16322853